CLINICAL TRIAL: NCT03934372
Title: An Open-Label, Single-Arm, Phase 1/2 Study Evaluating the Safety and Efficacy of Ponatinib for the Treatment of Recurrent or Refractory Leukemias, Lymphomas or Solid Tumors in Pediatric Participants
Brief Title: Safety and Efficacy of Ponatinib for Treatment of Pediatric Recurrent or Refractory Leukemias, Lymphomas or Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 84344-102; 2023-509699-41-00 (Registry Identifier: EU CT Number); 2018-004878-99 (EudraCT Number)
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Accelerated Phase Chronic Myeloid Leukemia; Blast Phase Chronic Myeloid Leukemia; Chronic Phase Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia; Leukemia; Lymphoma; Solid Tumors
Keywords: Leukemia; Solid tumors; Pediatric; Tyrosine kinase inhibitor; lymphomas
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphoma | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ponatinib (Experimental): Phase 1: Ponatinib administered according to age-based cohort doses and formulations to determine the maximum tolerated dose and recommended Phase 2 dose. Phase 2: Ponatinib administered at the recommended Phase 2 dose.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib administered as a tablet or age-appropriate formulation for pediatric participants according to age-based cohort assignment.
  Other Names: Iclusig, INCB84344

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and efficacy of ponatinib in children aged 1 to < 18 years with advanced leukemias, lymphomas, and solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed diagnosis of the following malignancies:

- Phase 1: CP-CML, BP-CML, AP-CML ALL. AML. Other leukemias. Lymphoma. Any other tumors, including tumors of the CNS, for which standard therapy is not available or is not indicated.

- Phase 2, Group A with CP-CML: CP-CML at the time of study entry and must be resistant to or intolerant of at least 1 prior BCR-ABL-targeted TKI therapy or be in "warning" response status or have the T315I kinase domain mutation.

Must have 1 bone marrow aspirate with documentation of BCR-ABL translocation by conventional cytogenetics, metaphase FISH, or q-PCR performed within 42 days before the first dose of ponatinib.

- Phase 2, Group B with other leukemias or solid tumors: ALL. AML. Other leukemias. Lymphoma. Any other tumors, including tumors of the CNS, with mutations of RET, FLT3, KIT, FGFR, PDGFR, TIE2, VEGFR, or any other mutations where ponatinib may have biological activity (eg, EPH receptors and SRC families of kinases) as assessed on fresh or archived tumor tissue.

Participants with solid tumors or with lymphoma must have measurable disease by CT or MRI based on RECIST v1.1 or the Lugano lymphoma guidelines as determined by site radiology.

Prior therapies as follows:

- Phase 1: Participants with CML who are resistant to or intolerant of (as defined Appendix F) to at least 1 prior BCR-ABL-targeted TKI therapy.

Participants with ALL who have progressed on or after all available or indicated therapies, which may have included 1 prior BCR-ABL-targeted TKI therapy.

Participants with AML or other leukemias who have progressed on or after at least 1 prior induction attempt (for France only) or for whom no effective standard therapy is available or indicated (other countries).

Participants with solid tumors (including tumors of the CNS) or lymphomas who have progressed despite standard therapy or for whom no effective standard therapy is available or indicated.

- Phase 2, Group A with CP-CML: Participants who are resistant to or intolerant of at least 1 prior BCR-ABL-targeted TKI therapy.

- Phase 2, Group B with other leukemias or solid tumors: Participants with ALL who have progressed on or after all available or indicated therapies, which must have included 1 prior BCR-ABL-targeted TKI therapy.

Participants with AML or other leukemias who have progressed on or after at least 1 prior induction attempt (for France only) or for whom no effective standard therapy is available or indicated (other countries).

Participants with solid tumors (including tumors of the CNS) or lymphomas who progressed despite standard therapy or for whom no effective standard therapy is available or indicated.

* Karnofsky performance status ≥ 40% for participants ≥ 16 years old or Lansky Play Scale ≥ 40% for pediatric participants < 16 years old.
* Participants must have recovered to < Grade 2 per the NCI CTCAE v5.0 or to baseline from any non-hematologic toxicities (except alopecia) due to previous therapy.
* Willingness to avoid pregnancy or fathering children.

Prior therapies:

- Participants with BP-CML, ALL, or AML who have received any of the following: Corticosteroids or hydroxyurea within 24 hours before the first dose of ponatinib.

Vincristine within 7 days before the first dose of ponatinib. Other chemotherapy (excluding intrathecal chemotherapy) within 14 days before the first dose of ponatinib.

- Participants (except the BP-CML, ALL, and AML participants described above) who: Have had cytotoxic chemotherapy within 21 days (or 42 days for nitrosoureas or mitomycin C) before the first dose of ponatinib.

Prior radiation therapy or radio-isotope therapy within 6 weeks before the first dose of ponatinib except local radiotherapy for palliative indication within 14 days before the first dose of ponatinib.

Autologous or allogeneic stem cell transplant < 3 months before the first dose of ponatinib.

Major surgery within 14 days before the first dose of ponatinib. Inadequate recovery and/or complications from a major surgery before starting therapy.

Prior treatment with any of the following:

* Immunosuppressive therapy (including post stem cell transplant regimens) within 14 days before the first dose of ponatinib.
* Any targeted cancer therapy (including TKIs) within 7 days before the first dose of ponatinib.
* Any other investigational anticancer agents within 30 days or 5 half-lives, whichever is longer, before randomization.
* Any monoclonal antibody-directed anticancer therapy within 5 half-lives of the first dose of ponatinib.
* Any chimeric antigen receptor therapy within 28 days before the first dose of ponatinib
* Ponatinib
* Protocol-defined lab Values
* Significant concurrent, uncontrolled medical condition, including but not limited to the following:
* Pancreatic: clinical, radiological, or laboratory evidence of pancreatitis.
* Cardiac:
* SF < 27% by ECHO, OR EF < 50% by MUGA.
* Abnormal QTcF on screening ECG, defined as QTcF of ≥ 450 ms.
* Clinically significant or uncontrolled cardiovascular disease, including unstable angina, acute MI within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV CHF (see Appendix P), and arrhythmia requiring therapy unless approved by the medical monitor/sponsor.
* Uncontrolled hypertension.
* Currently taking drug(s) that are known to have a risk of causing prolonged QTc or TdP unless the drug(s) can be changed to acceptable alternatives (ie, an alternate class of agents that do not affect the cardiac conduction system), or the participant can safely discontinue the drug(s).
* Cerebral:
* Participants with solid tumors with intracranial metastasis OR participants with active CNS leukemia (ie, CNS-2 status [< 5/μL WBCs and cytospin positive for blasts, or ≥ 5 /μL WBCs but negative by Steinherz/Bleyer algorithm (equation used for traumatic lumbar punctures), disseminated leptomeningeal disease, or CNS chloroma.
* Pre-existing significant CNS pathology including history of severe brain injury, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination/movement disorder, or autoimmune disease with CNS involvement.
* History of cerebrovascular ischemia/hemorrhage with residual deficits.
* Note: Participants with a history of cerebrovascular ischemia/hemorrhage remain eligible provided all neurologic deficits have resolved clinically according to Inclusion Criterion 6.
* Uncontrolled seizure disorder.
* Coagulation:
* Significant bleeding disorder or thrombophilia unrelated to the underlying malignancy indication for study participation.
* Gastrointestinal:
* Gastrointestinal disorders, such as malabsorption syndrome or any other illness that could affect oral absorption.
* Genetic:
* Participants with DNA fragility syndromes, such as Fanconi anemia and Bloom syndrome.
* Participants with Down syndrome.
* Participants with any active ≥ Grade 2 graft versus host disease.
* Chronic or current active uncontrolled infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment.
* Active HBV or HCV infection that requires treatment or at risk for HBV reactivation. Hepatitis B virus DNA and HCV RNA must be undetectable upon testing. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive.
* Known HIV infection.
* Current use of prohibited medication (see Section 6.7.2).
* Known hypersensitivity or severe reaction to ponatinib or excipients of ponatinib.
* Receipt of live (including attenuated) vaccines or anticipation of need for such vaccines during the study.
* Inability or unlikeliness to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* Females who are pregnant or lactating.
* Other exclusions may apply.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of dose-limiting toxicities | 28 days
  Defined as the occurrence of any protocol-defined toxicities occurring after dosing and up to and including Day 28, except those toxicities with a clear alternative explanation.
Phase 2: Efficacy of ponatinib assessed by major cytogenetic response (MCyR) in participants with chronic-phase chronic myeloid leukemia (CP-CML) | 12 months
  Defined as complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR) as assessed by conventional cytogenetics or fluorescence in situ hybridization (FISH).
Phase 2: Efficacy of ponatinib assessed by major hematologic response (MaHR) or major molecular response (MMR) in participants with BCR-ABL-positive leukemias | 3 months
  Assessed by polymerase chain reaction (PCR).
Phase 2: Efficacy of ponatinib assessed by complete response (CR) in participants with leukemias other than BCR-ABL-positive leukemias to determine the efficacy of ponatinib | 6 months
Phase 2: Efficacy of ponatinib assessed by incomplete complete response (iCR) in participants with leukemias other than BCR-ABL-positive leukemias | 6 months
  Assessed by conventional cytogenetics, FISH, or PCR.
Phase 2: Efficacy of ponatinib assessed by CR in participants with lymphoma | 6 months
  According to Lugano criteria based on computed tomography (CT) or magnetic resonance imaging (MRI) (or positron emission tomography [PET]).
Phase 2: Efficacy of ponatinib assessed by overall response rate in participants with solid tumors | 6 months
  Defined as the percentage of participants having CR or PR, as determined by investigator assessment of radiographic disease per tumors per RANO for central nervous system (CNS) tumors or Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) for other solid tumors based on CT or MRI (or PET).

SECONDARY OUTCOMES:
Phase 1: Number of treatment-emergent adverse events | 6 months
Phase 1: Tmax of ponatinib | 6 months
  Time to maximum concentration.
Phase 1: AUCss,0-24 of ponatinib | 6 months
  Area under the steady-state plasma or serum concentration-time curve from Hour 0 to 24.
Phase 1: t½ of ponatinib | 6 months
  Apparent terminal-phase disposition half-life.
Phase 1: CLss/F of ponatinib | 6 months
  Apparent oral dose clearance at steady state.
Phase 1: Vz/F of ponatinib | 6 months
  Apparent oral dose volume of distribution.
Phase 1: MCyR in participants with BCR-ABL-positive leukemias | 3 months
  Defined as CCyR or PCyR as assessed by conventional cytogenetics or FISH.
Phase 1: MMR in participants with BCR-ABL-positive leukemias | 3 months
  Assessed by quantitative PCR (q-PCR).
Phase 1 and Phase 2: Complete hematologic response (CHR) in participants with CP-CML | 6 months
Phase 1 and Phase 2: CCyR in participants with CP-CML | 12 months
Phase 1 and Phase 2: MMR in participants with CP-CML | 12 months
Phase 1 and Phase 2: Time to response (TTR) in participants with CP-CML | 6 months
  Defined as the interval from the date of the first dose of study treatment to first response.
Phase 1 and Phase 2: Duration of response (DOR) in participants with CP-CML | 6 months
  Defined as the interval between the first assessment at which the criteria for response are met until the criteria for progression are met.
Phase 1 and Phase 2: Progression-free survival (PFS) in participants with CP-CML | 6 months
  Defined as the interval from the date of the first dose of study treatment until the date of progression of disease or the date of death from any cause, whichever is earlier.
Phase 1 and Phase 2: Overall survival (OS) in participants with CP-CML | 6 months
  Defined as the interval from the date of the first dose of study treatment until death from any cause.
Phase 1: CR in participants with leukemias other than BCR-ABL-positive leukemia or CP-CML. | 6 months
Phase 1: CRi in participants with leukemias other than BCR-ABL-positive leukemia or CP-CML | 6 months
  Assessed by conventional cytogenetics, FISH, or q-PCR.
Phase 1: CR in participants with lymphoma | 6 months
  According to Lugano criteria based on CT or MRI (or PET).
Phase 1: Overall response rate in participants with solid tumors | 6 months
  Defined as the percentage of participants having CR or PR, as determined by investigator assessment of radiographic disease per tumors per RANO for CNS tumors or RECIST v1.1 for other solid tumors based on CT or MRI (or PET).
Phase 2: Anticancer activity of ponatinib assessed by MaHR or MMR in participants with BCR-ABL-positive leukemias (AP-CML, BP-CML or Ph+ALL) | 3 months
Phase 2: Anticancer activity of ponatinib assessed by CR in participants with leukemias other than BCR-ABL-positive leukemias | 6 months
Phase 2: Anticancer activity of ponatinib assessed by CRi in participants with leukemias other than BCR-ABL-positive leukemias. | 6 months
  Assessed by conventional cytogenetics, FISH, or PCR.
Phase 2: Anticancer activity of ponatinib assessed by CR in participants with lymphoma | 6 months
  According to Lugano criteria based on CT or MRI (or PET).
Phase 2: Anticancer activity of ponatinib assessed by overall response rate in participants with solid tumors | 6 months
  Defined as the percentage of participants having CR or PR, as determined by investigator assessment of radiographic disease per tumors per RANO for CNS tumors or RECIST v1.1 for other solid tumors based on CT or MRI (or PET).
Phase 2: OS in participants with solid tumors | 6 months
  Defined as the interval from the date of the first dose of study treatment until death from any cause.
Phase 2: DOR in participants with solid tumors | 6 months
  Defined as the interval between the first assessment at which the criteria for response are met until the criteria for progression are met.
Phase 2: PFS in participants with solid tumors | 6 months
  Defined as the interval from the date of the first dose of study treatment until the date of progression of disease or the date of death from any cause, whichever is earlier.
Phase 2: Number of treatment-emergent adverse events | 6 months
Phase 2: Clearance of pediatric-friendly formulation of ponatinib | 6 months
Phase 2: Volume of distribution of pediatric-friendly formulation of ponatinib | 6 months
Phase 2: AUC of pediatric-friendly formulation of ponatinib | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed-El-Amine Bensmaine, MD, Study Director — Incyte Biosciences International Sàrl
Locations (25):
- Ghent University Hospital, Ghent, Belgium
- France (4):
  - Hopital Robert Debre, Paris
  - Armand Trousseau Hospital, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Chu de Rennes - Hospital Sud, Rennes
- Italy (9):
  - Aou Policlinico S. Orsola-Malpighi, Bologna
  - Asst Degli Spedali Civili Di Brescia, Brescia
  - Ospedale Pediatrico G. Gaslini, Genova
  - Comitato Etico Fondazione Irccs Istituto Nazionale Dei Tumori Milano, Milan
  - University of Milano Bicocca, Monza
  - Aorn Santobono Pausilipon, Naples
  - Comitato Di Bioetica Della Fondazione Irccs Policlinico San Matteo, Pavia
  - Ospedale Pediatrico Bambino Gesu Irccs, Rome
  - A.O.U Citta Della Salute E Della Scienza Di Torino Presidio Ospedaliero Infantile Regina Margherita, Torino
- Princess Maxima Center For Pediatric Oncology, Utrecht, Netherlands
- Spain (4):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Sant Joan de Deu de Manresa, Barcelona
  - Hospital Infantil Unversitario Nino Jesus, Madrid
  - Hospital Universitari I Politecnic La Fe, Valencia
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna, Solna
  - Karolinska University Hospital Solna, Stockholm
- United Kingdom (4):
  - Royal Hospital For Sick Children Yorkhill Glasgow, Glasgow
  - Alder Hey Childrens Nhs Foundation Trust, Liverpool
  - The Royal Marsden Nhs Foundation Trust - Sutton, Sutton
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Safety and Efficacy of Ponatinib for Treatment of Pediatric Recurrent or Refractory Leukemias, Lymphomas or Solid Tumors — https://incyteclinicaltrials.com/studies/incb-84344-102